CLINICAL TRIAL: NCT04815447
Title: Cardiopulmonary Fitness and Its Clinical Determinants of a Population of Childhood Cancer Survivor: a Controlled Retrospective Study
Brief Title: Cardiopulmonary Fitness and Its Clinical Determinants of a Population of Childhood Cancer Survivor
Acronym: ONCO-SPORT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Pediatric Oncology Department, Montpellier University Hospital, France (Unknown); Pediatric and Congenital Cardiology Department, Montpellier University Hospital, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0089
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Childhood Cancer
Keywords: childhood cancer survivors; VO2max; Ventilatory anaerobis threshold; Cardio-pulmonary exercise test; Hematopoietic stem cells transplantation; Radiotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CCS group: Patients under 25 were recruited in the pediatric CPET laboratory of Montpellier University Hospital after a regular paediatric cardiology outpatient visit.
- Control: The control group consisted in children referred for a non-severe functional symptom linked to exercise (murmur, palpitation, or dyspnoea) or for a medical sports certificate. These children were classified in the control group only after a completely normal check-up, including physical examination, electrocardiogram, echocardiography, and spirometry.

SUMMARY:
Medical progress have made it possible to considerably improve the survival of children with an oncological disease. Currently, the survival rate increased to above 90 % in the most developed countries . This increase of childhood cancer survivors (CCS) asks us about their future and their quality of life. Assessing health related life quality , previous studies observe that in this particular population of patients, it is related to a poor physical capacity , physical activity level and many of these patients do not meet the activity level recommended by the world health organization due to fatigability and sedentary behaviours . In addition to these habits, the CCS are more susceptible to develop cardiovascular risk (CVR) leading to cardiovascular disease in adulthood and increases them mortality . Furthermore, CCS who have been experiencing hematopoietic stem cells transplantation (HSCT) are more susceptible to develop these CVR. In parallel with the common CVR, lower cardiopulmonary fitness assessed by cardiopulmonary exercise test (CPET) in the general population has been established as a major and independent CVR for cardiologic events.

Cardiopulmonary fitness assessed by maximal cardiopulmonary exercise test (CPET) allows physicians to measure metabolic response to maximal effort in a population that is known as VO2max. This domain of applied physiology permits a new way to approach the understanding of global health prognosis in chronic disease. For example, decrease of VO2max is involved in lower quality of life in patients with congenital heart disease. Cardiopulmonary exercise test for VO2max exploration has been demonstrated feasible in child patients with leukemia or other tumors after intensive chemotherapy, prior to HSCT.

Assessment of cardiopulmonary fitness in CCS is already described in previous studies, but this study aimed to compare a maximal CPET assessment on a large childhood cancer survivors cohort with healthy control, on a quite young cohort, during the oncologic follow up and find out its determinants.

DETAILED DESCRIPTION:
This is a controlled, monocentric, cross-sectional study conducted in a tertiary care center for oncologic disease in children (Montpellier University Hospital, France) was carried out between November 2010 and November 2020.

Two groups were identified: CCS group and control group.

ELIGIBILITY:
Inclusion criteria for CCS group :

* aged between 5 and 25 years old,
* having been complete a full regimen for oncological disease and considered in remission at the end of treatment. Remission was considered in absence of relapse or new treatment initiated before the CPET end point.

Inclusion criteria for control group :

* children referred for a nonsevere functional symptom linked to exercise (murmur, palpitation or dyspnoea) or for a medical sports certificate.
* completely normal check-up, including physical examination, ECG, echocardiography and spirometry.

Exclusion criteria for control group:

* Children with any chronic disease, medical condition (cardiac, neurological, respiratory, muscular or renal)
* Children with any medical treatment
* Children requiring any further specialised medical consultation

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * CCS having been complete a full regimen for oncological disease and considered in remission at the end of treatment
  * Controlled children with completely normal check-up, including physical examination, ECG, echocardiography and spirometry
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
comparison of VO2max for CCS patients compared to control children | 1 day
  comparison of the mean of VO2max value in ml/kg/min between CCS group and control group

SECONDARY OUTCOMES:
comparison of ventilatory anaerobic threshold (VAT) for CCS patients compared to control children | 1 day
  comparison of the mean of VAT value in ml/kg/min between CCS group and control group
correlation between clinical determinants and VO2max in the CCS group | 1 day
  with multivariate analysis, we will look for the correlation between the clinical determinants and the decreased of VO2max in CCS group.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD, PhD, Study Director — University Hospital, Montpellier; Arthur GAVOTTO, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Gavotto A, Dubard V, Avesani M, Huguet H, Picot MC, Abassi H, Guillaumont S, De La Villeon G, Haouy S, Sirvent N, Sirvent A, Theron A, Requirand A, Matecki S, Amedro P. Impaired aerobic capacity in adolescents and young adults after treatment for cancer or non-malignant haematological disease. Pediatr Res. 2023 Aug;94(2):626-631. doi: 10.1038/s41390-023-02477-6. Epub 2023 Jan 28. PMID 36709386